CLINICAL TRIAL: NCT05582317
Title: Efficacy of Combination of Biodentine and Simvastatin as a Pulp Capping Materials in Vital Pulpotomy of Primary Molars: - a Clinical and Experimental Study
Brief Title: Efficacy of Combination of Biodentine and Simvastatin as a Pulp Capping Materials in Vital Pulpotomy of Primary Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-293
Record Dates: First submitted 2022-09-12; First posted 2022-10-17 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-08

CONDITIONS: Pulpitis - Irreversible
MeSH Terms: interventions — tricalcium silicate; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Biodentine (Active Comparator): 20 primary molars were treated by Biodentine
  Interventions: Drug: Biodentine
- Simvastatin (Active Comparator): 20 primary molars were treated by Biodentine
  Interventions: Drug: Simvastatin
- combination of Biodentine and Simvastatin (Active Comparator): 20 primary molars were treated by Biodentine
  Interventions: Drug: Biodentine; Drug: Simvastatin

INTERVENTIONS:
Drug: Biodentine — Tricalcium silicate, dicalcium silicate, calcium carbonate and oxide filler, iron oxide shade and zirconium oxide
  Arms: Biodentine; combination of Biodentine and Simvastatin
Drug: Simvastatin — 3-hydroxy-3-methylglutaryl coenzyme A reductase inhibitor
  Arms: Simvastatin; combination of Biodentine and Simvastatin

SUMMARY:
Objective: This study was conducted to evaluate the efficacy of combination of biodentine with simvastatin as a pulpotomy agent for vital primary molars clinically and radiographically.

Study design: 60 primary molars in 20 children aged 4-7 years old were randomly allocated to three groups, Biodentine, Simvastatin and combination of Biodentine and simvastatin. Clinical and radiographic examinations were conducted at 1, 3, 6, 9 and 12 months after treatment.

Key words: Pulpotomy, Primary teeth, Biodentine, Simvastatin.

DETAILED DESCRIPTION:
Each tooth will be locally anesthetized using topical anesthetic gel benzocaine 20% on the mucosa after drying the area with gauze; the application of local anesthesia using Mepivacaine Hydrocholride 2% with Levonordefrin 1:20000 to the tooth following the recommended technique for each tooth to be treated; then the tooth will be isolated using rubber dam and high suction 3. The pulpotomy procedures will be performed as follow:- All soft caries will be removed by large spoon excavator. Cavity outline will be performed using a sterile #330 carbide bur at high speed (30,000 rpm) contra-angle hand piece will be used under a water coolant.

* Access to a pulp chamber will be detected with a probe, or if the roof of the pulp chamber is sufficiently thin to see the pulpal tissue. When the pulpal exposure is confirmed, the roof of the pulp chamber will be removed with a sterile large low speed round bur #4 with water spray.
* The coronal pulp will be amputated using a sterile sharp spoon excavator, until the orifices of the stumps can be seen clearly without remnant tags and the access will be refined with a sterile high speed fissure bur (El sayed et al., 2019).
* The pulp chamber will be irrigated with normal saline.
* Pulp hemostasis will be achieved using a wet cotton pellet with sterile saline applied on the radicular pulp stumps under slight pressure for 2 to 3 minutes.
* If bleeding cant be controlled within 5 minutes, the tooth will be excluded from the study and the needed treatment will be done.

  4. Depending on group allocation, the pulp stumps of molars will be dressed as follows:

Group (I): 20 primary molars were treated with Biodentine :-

The mixture of Biodentine will be made according to manufacturer's directions as follow:

i. Biodentine is available in the form of a pre-measured capsule and a liquid in a pipette ii. Before the Biodentine capsule is opened, it is tapped gently on a hard surface to diffuse the powder.

iii. Five drops of liquid from the single-dose dispenser is poured into the capsule, then it is placed in an amalgamator and mixed for 30 sec .

iv. The mixture is recovered with the aid of the manufacturer supplied spatula.

* The mixture of Biodentine is introduced into the pulp chamber using amalgam carrier, uniformly placed over the floor of pulp chamber and compacted with a condenser

Group (II):20 primary molars were treated with Simvastatin :-

* Simvastatin powder 1.5 mg is mixed with distilled water to get homogenous paste (Shaheen et al., 2018)
* The mixture of Simvastatin then iss delivered to into the pulp chamber using a plastic instrument and compacted with a condenser

Group (III): 20 primary molars isre treated with combination of Biodentine and Simvastatin:-

• 1:1 of mixture of Biodentine and Simvastatin paste, using one measurable instrument, they will be together and the mixture will be delivered to into the pulp chamber using a plastic instrument and compacted with a condenser

5. In three groups the access cavity of all treated molars is filled by restorative glass ionomer cement and all molars are finally restored with stainless steel crowns and cemented by glass ionomer cement

6. Post-operative digital radiograph will be taken at the same visit for all treated primary molars (0-baseline) 7. The patients is instructed to perform oral hygiene measures (teeth brushing twice daily) under supervision of their parents.

8. Clinical follow up will be done after (one, three, six, nine and twelve) months.

Digital Radiographic follow up will be done after (three, six, nine and twelve) months.

Radiographic examination: It will be done by taking aiagnostic pre-operative digital periapical radiograph using size 0 Phosphostimulable Phosphor plates (PSP), scanner and x-ray machine at Oral Radiology Department ,Faculty of Dentistry ,Suez Canal University to assess the inclusion and exclusion criteria.

9. The patient is asked to come to the clinic between follow up visits if he/she has any complain from the treatment, and the alternative treatment will be done according to the case.

A.II.7: Methods of Evaluation:

The pulpotomized teeth are judged as clinically and radiographically successful if they met the following criteria (Elbardissy et al., 2019).

Clinically:

Absence of pain. No tender on percussion. No swelling/sinus. No pathological tooth mobility.

Radiographically:

No loss of lamina dura. Normal periodontal ligament space. No external/internal resorption. No periapical /furcation radiolucency. Evaluation will be done by two independent evaluators Treatment is considered as clinically failure when one or more of the following signs (pain, tender on percussion swelling/sinus or pathological tooth mobility) were detected and radiographically failure when one or more of the following signs (lamina dura, widening in periodontal ligament space presence of external/internal resorption or presence of periapical /furcation radiolucency) were detected . Time for teeth with pulpotomy failure was defined as the time elapsed between treatment and the first visit in which pathologic finding was detected. When failure was detected, the tooth was traditionally treated with zinc oxide eugenol pulpectomy or extracted and excluded from the study

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy children free from any known systemic diseases.
* Parent willing to participate in the study and signed an informed consent.
* Patient had at least three restorable primary molars with a caries- exposed vital pulp

Exclusion Criteria:

* history of spontaneous pain or provoked pain.
* clinical signs and ̸ or symptoms suggesting a non-vital tooth such as (fistula, sinus tract, soft tissue swelling, mobility or tenderness to percussion).
* non-Restorable tooth
* pathologic or physiologic mobility

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2021-05-23 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
Clinical assessment | 12 months
  Pain, tenderness, Swelling No tender on percussion. No swelling/sinus. No pathological tooth mobility.

SECONDARY OUTCOMES:
Radiographically: | 12 months
  Lamina dura, periodontal ligament space, resorption Normal periodontal ligament space. No external/internal resorption. No periapical /furcation radiolucency.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, Suez canal university, Ismailia, Egypt